CLINICAL TRIAL: NCT00577304
Title: A Study of a Topical Formulation of Nitroglycerin, MQX-503, and Matching Vehicle in the Treatment and Prevention of Raynaud's Phenomenon
Brief Title: A Study of a Topical Form of Nitroglycerin and Placebo in the Treatment and Prevention of Raynaud's Phenomenon
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MediQuest Therapeutics (Industry)
Responsible Party: Fred Dechow/President and CEO, MediQuest Therapeutics, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-005
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2008-04

CONDITIONS: Raynaud's Disease; Raynaud's Disease Secondary to Scleroderma; Raynaud's Disease Secondary to Other Autoimmune Disease
Keywords: Raynaud's; Nitroglycerin; Scleroderma
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Diffuse | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Other): Placebo - Topical AmphiMatrix
  Interventions: Drug: Topical AmphiMatrix
- 1 (Active Comparator): Topical AmphiMatrix with Nitroglycerin
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Nitroglycerin — Individual pouch applicators containing 0.5 grams of Topical AmphiMatrix with Nitroglycerin. Each dose contains 4.5mg of Nitroglycerin. Each dose is intended for topical usage on both hands up to five minutes before an anticipated Raynaud's attack or up to 5 minutes after the beginning of an actual Raynaud's attack. Limited to four applications per day; minimum of two hours between applications.
  Arms: 1
Drug: Topical AmphiMatrix — Individual pouch applicators containing 0.5 grams of Topical AmphiMatrix. Each dose is intended for topical usage on both hands up to five minutes before an anticipated Raynaud's attack or up to 5 minutes after the beginning of an actual Raynaud's attack. Limited to four applications per day; minimum of two hours between applications.
  Arms: 2

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of Topical AmphiMatrix with Nitroglycerin (MQX0503) to relieve Raynaud's symptoms and increase blood flow to the fingers.

DETAILED DESCRIPTION:
The purpose of this clinical study is to determine, in a controlled fashion, the ability of a topical formulation of Nitroglycerin, MQX-503, to improve the patient's health assessment as indicated by patient and physician assessments, decrease the frequency of Raynaud's events, decrease the duration of Raynaud's events, and decrease the symptoms (pain, tingling, numbness) in the fingers of Raynaud's patients. The study will include patients with moderate to severe primary Raynaud's Phenomenon (RP) and with moderate to severe Raynaud's Phenomenon secondary to autoimmune diseases, such as scleroderma.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ages 15 - 70.
* Patients with a diagnosis of Raynaud's phenomenon.
* Patients who agree to apply study medication to their fingers.
* Patients who are willing to stop current topical vasodilator therapies.
* Patients who agree not to start or change dosage of current oral vasodilator therapies.
* Patients who agree not to use any nitrate therapy while participating in this study.
* Negative pregnancy test in fertile women and agreement to use effective contraception throughout the study.

Exclusion Criteria:

* Patients who currently use nitrate medication or medications known to interact with nitroglycerin.
* Patients who have an allergy to nitroglycerin or common topical gel ingredients.
* Patients with a history of severe headaches.
* Patients with an unstable medical problem.
* Patients with cognitive or language difficulties that would impair their ability to complete assessment of pain instruments.
* Patients who have had a recent heart attack or other uncontrolled heart condition.
* Patients who have participated in an investigational drug study within four weeks of visit one.
* Patients who have clinically significant abnormal lab values.
* Patients who have had recent major abdominal, thoracic or vascular surgery.
* Patients with interfering skin conditions.
* Pregnant or nursing women or women unwilling to comply with contraceptive requirements.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-03 (Estimated); Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in Raynaud's Condition Score | three months

SECONDARY OUTCOMES:
Frequency and severity of adverse events. | three months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Ohrstrom, PhD, Study Director — MediQuest Therapeutics
Locations (17):
- United States (17):
  - Stanford University, Stanford, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Arthritis Education and Treatment Center, PLLC, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - The Center for Rheumatology, Albany, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Carolina Arthritis, Wilmington, North Carolina
  - University of Toledo, Toledo, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas at Houston, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Sponsor web site — http://www.mqti.com